CLINICAL TRIAL: NCT06066671
Title: Evaluation of the Effect of na Experimental Gel Based on Copaiba Oil Resin in Reducing Post-bleaching Tooth Sensitivity: a Randomized Clinical Study
Brief Title: The Effect of an Experimental Gel Based on Copaiba Oil Resin in Reducing Post-bleaching Tooth Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Professor of the graduate program in dentistry at Federal Univeersity of Pará, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara016
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Tooth Bleaching Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GCO (Experimental copaiba oil resin gel) (Experimental): The GCO group will receive the application of an experimental gel based on copaiba oil resin for post tooth bleaching sensitivity
  Interventions: Other: GCO (Experimental copaiba oil resin gel)
- GN (Potassiun nitrate and sodium fluoride gel) (Active Comparator): The GN group will receive the application of a potassium and sodium nitrate gel for post tooth bleaching sensitivity
  Interventions: Other: GCO (Experimental copaiba oil resin gel)
- GC (Placebo Comparator): The GC group will receive the application of a placebo gel for post tooth bleaching sensitivity
  Interventions: Other: GCO (Experimental copaiba oil resin gel)

INTERVENTIONS:
Other: GCO (Experimental copaiba oil resin gel) — Prior to bleaching treatment with 35% hydrogen peroxide, the dental elements of the GCO will receive the application of the experimental desensitizing gel on the buccal surfaces of the central incisors, lateral incisors, canines and upper and lower premolars, with a rubber cup in an active way, for 10 minutes.

SUMMARY:
This randomized, double-blind clinical trial aimed to evaluate the effect of an experimental gel containing copaiba oil resin in reducing postoperative tooth sensitivity caused by bleaching with 35% hydrogen peroxide. The volunteers of this study were randomized into 3 different groups - GC (placebo); GN (potassium nitrate and sodium fluoride); GCO (copaiba oil resin). The dental elements of the GCO received application of the experimental desensitizing gel on the buccal surfaces of the central incisors, lateral incisors, canines and upper and lower premolars, with a rubber cup in an active way, for 10 minutes. The GC and GN groups also received the application of a placebo gel and a nitrate potassium and sodiun fluoride gel, respectively, under the same conditions described for the experimental gel. Subsequently, all groups underwent in-office bleaching treatment with 35% hydrogen peroxide. Post-bleaching sensitivity was collected through a form composed of the visual analogue scale (VAS). Color measurement was performed at two times: baseline (Ti) and one week after the 3rd bleaching session (Tf).

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene
* absence of active caries lesions
* never undergone bleaching therapy
* not present dental hypersensitivity
* don't be a smoker
* don´t be pregnant
* present at least 28 teeth in the oral cavity

Exclusion Criteria:

* volunteers undergoing orthodontic treatment,
* presence of periodontal disease
* dental cracks or fractures
* restorations and prostheses on anterior teeth
* extensive molar restorations
* gastroesophageal disorders
* severe internal dental darkening
* presence of dentinal exposure in anterior and / or posterior teeth.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Assessment of post-bleaching sensitivity | 21 days
  For the assessment of postoperative sensitivity, patients were instructed to fill out a form to record tooth sensitivity daily, during the 21 days of treatment, based on individual pain perception. This form was delivered at each bleaching session, being returned to the researcher in the following session, that is, always one week after each bleaching session. The evaluation form consisted of the visual analogue scale (VAS). This scale consists of a 10 cm horizontal line, with scores of 0 and 10 at its ends, where 0 means no sensitivity and 10 means severe tooth sensitivity. The patient was instructed to draw a vertical line along the horizontal line of the scale, recording the intensity of tooth sensitivity per day. So that the distance in millimeters from the zero end could be later measured with the aid of amillimeter ruler, thus obtaining the patient's level of pain intensity.

SECONDARY OUTCOMES:
Color evaluation | Baseline (Ti) and one week after the 3rd bleaching session (Tf)
  The VITA Easyshade spectrophotometer (VITA Zahnfabrik, Bad Säckingen, Germany) was used to measure the color, where the area of dental correspondence to be evaluated was the middle third of the buccal surface of the upper canines. To standardize the color readings, silicone trays were made, where the impression was extended from canine to canine. A window was created on the buccal surface of each canine of the silicone guide using a metal device with a 6 mm radius, corresponding to the diameter of the spectrophotometer tip. Thus, the tip of the device was inserted into the silicone guide to obtain the color parameters. Subsequently, the color difference between baseline (T i) and one week after the 3rd bleaching session (T f ) was calculated using the CIEDE2000 formulas (ΔE00).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Para, Belém, Pará, Brazil